CLINICAL TRIAL: NCT04473131
Title: Immune Profiling of COVID-19-infected Patients Admitted to the Intensive Care Unit (ICU): the IMPROVISE Study
Brief Title: Immune Profiling of COVID19-patients Admitted to ICU
Acronym: IMPROVISE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hamad Medical Corporation (Industry)
Collaborators: Qatar University (Other); Weill Cornell Medical College in Qatar (Other)
Responsible Party: Principal Investigator, Ali Ait Hssain, Senior consultant intensivist, Hamad Medical Corporation
Other Study IDs: MRC-05-007
Record Dates: First submitted 2020-07-15; First posted 2020-07-16 (Actual); Last update posted 2020-07-16 (Actual); Status verified 2020-07

CONDITIONS: COVID-19
Keywords: COVID-19; SARS-CoV-2; ICU; Immune profiling; Humoral immunity; Cellular immunity
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — EDTA blood samples Yellow SST blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- COVID-19 positive: Inclusion criteria:
  1. Male or female aged over 18 years
  2. Admitted patients to ICU with a suspicious COVID19 infection
  3. Tested positive for SARS-CoV-2
  Exclusion criteria:
  1. Burn and trauma
  2. Any immunological diseases, or immunosuppressive medications
  3. Other immune-related conditions (cancer, hematological malignancies, bone marrow diseases or transplant)
  Sample collection time points: 4 to 5 (day 1-3, day 7, day 14, day 21, discharge day from ICU -between day 30-60- if possible)
  Interventions: Other: No intervention
- COVID-19 negative: Inclusion criteria:
  1. Male or female aged over 18 years
  2. Admitted patients to ICU
  3. Tested negative for SARS-CoV-2
  Exclusion criteria:
  1. Burn and trauma
  2. Any immunological diseases, or immunosuppressive medications
  3. Other immune-related conditions (cancer, hematological malignancies, bone marrow diseases or transplant)
  Sample collection time points: 4 to 5 (day 1-3, day 7, day 14, day 21, discharge day from ICU -between day 30-60- if possible)
  Interventions: Other: No intervention
- Heathy volunteers: Inclusion criteria:
  1. Male or female aged over 18 years
  2. Normal clinical examination
  Exclusion criteria:
  1. Person with an infectious syndrome during the last 90 days
  2. Extreme physical stress within the last week
  3. Person receiving within the last 90 days, a treatment based on: antivirals; antibiotics; antiparasitics; antifungals; non-steroidal anti-inflammatory drugs; immunosuppressive therapy; corticosteroids; therapeutic antibodies; chemotherapy
  4. Person with history of: innate or acquired immune deficiency; hematological disease; solid tumor; severe chronic disease; surgery or hospitalization within the last 2 years; pregnancy within the last year; participation to a phase I clinical assay during the last year; participation to a phase I clinical assay during the last year; pregnant or breastfeeding women; a person with restricted liberty or under legal protection
  Sample collection time points: 1 (day of blood sample donation)
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — Only blood samples will be taken from participants for this study

SUMMARY:
SARS-CoV-2 is the novel coronavirus responsible for COVID-19, coronavirus disease 2019. This new coronavirus was first detected in Wuhan, China in late December 2019. According to WHO, the incidence rate of COVID-19 is prominent among adults and elderly people, reaching so far >2 million cases globally. Meanwhile, confirmed death cases reached >126 thousands of reported cases in 185 countries and still increasing. We anticipate that immunological differences among COVID19-infected patients might be a reason behind the variation of patient outcomes. Therefore, we intend to investigate cellular and humoral immune responses of COVID19-positive patients, and we claim to discover new indicators of patients' prognosis. Our target population includes three categories of patients staying at ICU, HMC (COVID19-positive vs. COVID19-negative vs. healthy control). Throughout their ICU stay, multiple blood samples will be screened for leukocytes surface markers, leukocytes' production of certain molecules, and circulating cytokines/chemokines/checkpoint inhibitors. Their plasma/serum will be used as well for immune proteomics, metabolomics, and other serological tests. Such parameters can provide the more comprehensive status of COVID19-infected patients at infection onset, during treatment intake, and at recovery or relapse stage. Following analysis, the main prospective outcome of this study is to identify the most reflective markers of COVID19-positive patients' outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Admitted to ICU for suspicious COVID-19
* Signed consent form

Exclusion Criteria:

* Immuno-compromised or immuno-deficient patients
* Diagnosed with any immunological disorders, cancer, and onco-hematological diseases at the inclusion date
* Patients under treatment or treated within 5 years before inclusion or at the end of chemotherapy within the 6 months prior to inclusion date
* Patients under any immune-suppressive medications, antibody therapy, corticosteroids, bone marrow transplant under the last 6 months of inclusion
* Unsigned consent form

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: In this study, we are targeting to enroll two categories of patients from ICU: 100 COVID19-positive patients, and 100 COVID19-negative patients.
  In addition to 100 healthy volunteers from the blood donation center.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2020-04-27 (Actual); Primary Completion 2022-06 (Estimated); Study Completion 2022-06 (Estimated)

PRIMARY OUTCOMES:
To create an immune profile for each COVID19-positive patient during their ICU stay | 8 to 12 months
  A descriptive analysis of the innate and adaptive immune cells (phenotypically and functionally), along with circulating pro- and anti-inflammatory cytokines, and the dynamic change of immune cells and cytokines throughout the first 4 weeks of the COVID-19 infection.
To correlate patients' immune profile to disease severity and patient's outcome | 4 to 6 months
  A correlative analysis of the immune cells and cytokines levels with the COVID-19 severity and with the patient's outcome following their stay at the ICU. An attempt to identify markers associated with the disease severity and predictive measures to the patient's outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- Hamad Medical Corporation, Doha, Qatar

REFERENCES:
- [Derived] Bradic M, Taleb S, Thomas B, Chidiac O, Robay A, Hassan N, Malek J, Ait Hssain A, Abi Khalil C. DNA methylation predicts the outcome of COVID-19 patients with acute respiratory distress syndrome. J Transl Med. 2022 Nov 12;20(1):526. doi: 10.1186/s12967-022-03737-5. PMID 36371196